CLINICAL TRIAL: NCT00775658
Title: Effect of Olopatadine Hydrochloride 0.2% Ophthalmic Solution on Epicutaneous Skin Prick Testing With Histamine and Saline
Brief Title: Olopatadine Eye Drops and Allergy Skin Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, John Michael Fahrenholz, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 071260
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis
Keywords: allergy; skin testing; eye drops; antihistamines
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Hypersensitivity | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- olopatadine then placebo (Active Comparator): participants received olopatadine 0.2% opthalmic solution 1 drop into each eye at the same time each day for 7 to 10 days followed by 7-10 day washout period. They then received a placebo, normal saline opthalmic solution 1 drop into each eye at the same time each day for 7-10 days
  Interventions: Drug: olopatadine; Drug: placebo
- placebo then olopatadine (Active Comparator): participants received olopatadine 0.2% opthalmic solution 1 drop into each eye at the same time each day for 7 to 10 days followed by 7-10 day washout period. They then received a placebo, normal saline opthalmic solution 1 drop into each eye at the same time each day for 7-10 days
  Interventions: Drug: olopatadine; Drug: placebo

INTERVENTIONS:
Drug: olopatadine — olopatadine 0.2% opthalmic solution 1 drop into each eye at the same time each day
Drug: placebo — placebo, normal saline opthalmic solution 1 drop into each eye at the same time each day

SUMMARY:
Use of olopatadine ophthalmic solution (eye drops) will decrease allergy skin test reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Healthy volunteers (no major illnesses or active symptoms)

Exclusion Criteria:

* Known allergy or hypersensitivity to the drugs or components
* Pregnant or nursing women
* Women wishing to become pregnant during the study's duration
* Use of topical or oral medications with antihistaminic activity for 14 days proceeding randomization
* Dermatographism as evidenced on skin testing on visit 1
* Chronic urticaria active within the past 6 months
* Severe hypertension
* Psychiatric diagnoses which could potentially affect medication compliance, such as schizophrenia or delusional disorders, as determined by the investigator obtaining informed consent and based on the subject's past medical history
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Asthma, Sinus and Allergy Program Research, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew prior to any study procedure: 1 had and upper respiratory infection, 1 required use of oral anti histamine and 1 was lost to follow up
Period: First Intervention
Arm/Group | Olopatadine Then Placebo | Placebo Then Olopatadine
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Olopatadine Then Placebo | Placebo Then Olopatadine
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes both groups of participants
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Area (cm2) of the Wheal Size in Histamine Skin Test Response During Treatment With Olopatadine Compared to Placebo.
Time Frame: at baseline and at return visit (between study day 7-10)
Measure: Mean (Standard Deviation); unit: cm2
Groups:
- Olopatadine: double blind crossover
Arm/Group | Olopatadine | Placebo
Number analyzed (Participants) | 21 | 21
cm2 | 0.461 (0.279) | 0.464 (0.254)
Statistical Analysis 1: Comparison: Olopatadine vs Placebo; Before the study, we determined that a sample size of 18 would be adequate to detect a 20% difference in wheal and flare areas with 80% power and a significance level of 0.05; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

2. Primary Outcome: The Difference in Area (cm2) of the Flare Size in Histamine Skin Test Response During Treatment With Olopatadine Compared to Placebo.
Time Frame: at baseline and at return visit (between study day 7-10)
Population: Sample size determined that 18 participants would provide 80% power to detect a 20% difference with a significance level of 0.05.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Olopatadine | Placebo
Number analyzed (Participants) | 21 | 21
cm2 | 6.95 (4.68) | 8.31 (3.98)
Statistical Analysis 1: Comparison: Olopatadine vs Placebo; Test type: Superiority — Sample size determined that 18 participants would provide 80% power to detect a 20% difference with a significance level of 0.05; p = 0.09, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Adverse Events Data was lost and is not reported
Arm/Group | Olopatadine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size and majority female patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No